CLINICAL TRIAL: NCT00005427
Title: Cohort Study of Respiratory Illness in Early Childhood
Status: Terminated | Type: Observational
Why Stopped: Not a clinical trial.
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4345; R03HL049896 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

SUMMARY:
To analyze previously collected data on respiratory illness in early childhood.

DETAILED DESCRIPTION:
BACKGROUND:

The study built on a previous study funded by the Health Effects Institute, a non-profit foundation jointly supported by the U.S. Environmental Protection Agency and vehicle manufacturers. The previous study was a prospective cohort study of nitrogen dioxide (NO2) exposure and respiratory symptoms and illnesses during the first 18 months of life. Between January, 1988 and June, 1990, 1,315 infants were enrolled and then followed with collection of daily respiratory symptom data and serial monitoring of NO2 concentrations in their homes. The full protocol was completed by 823 subjects and a total follow-up experience of over one-half million days was accumulated. Follow-up ended in December, 1991 and analyses related to the study's principal focus, the health effects of NO2, was completed during the fall of 1992.

DESIGN NARRATIVE:

The analyses were directed at the following: 1) Time spent in day-care and the incidence and severity of respiratory illnesses; 2) Breast-feeding and the incidence and severity of respiratory illnesses during the first six months of life; 3) Determinants of wheezing and wheezing illnesses; 4) Determinants of a physician-diagnosis of asthma; 5) Exposure to woodsmoke and incidence and severity of respiratory illnesses; 6) Household demographics, including ethnicity, and incidence and severity of respiratory illnesses; 7) Determinants of the duration of respiratory illnesses; 8) The validity of retrospective parental reports of respiratory illness; 9) Parental perceptions of the risks of indoor and outdoor air pollution; 10) Clinical findings on assessment of ill children in the community.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-03; Study Completion 1995-02

REFERENCES:
- [Background] Bosken CH, Hunt WC, Lambert WE, Samet JM. A parental history of asthma is a risk factor for wheezing and nonwheezing respiratory illnesses in infants younger than 18 months of age. Am J Respir Crit Care Med. 2000 Jun;161(6):1810-5. doi: 10.1164/ajrccm.161.6.9903030. PMID 10852749
- [Background] Cushing AH, Samet JM, Lambert WE, Skipper BJ, Hunt WC, Young SA, McLaren LC. Breastfeeding reduces risk of respiratory illness in infants. Am J Epidemiol. 1998 May 1;147(9):863-70. doi: 10.1093/oxfordjournals.aje.a009540. PMID 9583717